CLINICAL TRIAL: NCT00946907
Title: Benign Acute Pericarditis: Brief Versus Longer Treatment. Randomized, Multicentric, Double Blind, Non Inferiority Trial
Brief Title: Benign Acute Pericarditis: Brief Versus Longer Treatment Using Aspirin
Acronym: pericardite
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was suspended by principal investigator's decision. All the sites were not opened, and the recruitment was so slow.
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PERICARDITE
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Pericarditis
Keywords: acute pericarditis; treatment; recurrence
MeSH Terms: conditions — Pericarditis; Recurrence | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aspirin (Active Comparator)
  Interventions: Drug: Aspirin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aspirin — 3000mg/day of aspirin during the 4th first days and 2000mg/day of aspirin during the 17th following days
  Arms: aspirin
Drug: placebo — 3000mg/day of aspirin during the 4th first days and 2000mg/day of placebo during the 17th following days
  Arms: placebo

SUMMARY:
Treatment of pericarditis largely remains empirical due to the relative lack of randomized controlled trials. Nevertheless, some recommendations have been formulated to guide management and follow-up of acute pericarditis. Aspirin or an NSAID at medium to high dosages is the mainstay of treatment. Optimal length of treatment is not established.

PERICARDITE is a French multicentric placebo controlled double blind randomized trial assessing efficacy of a brief treatment based on Aspirin (4 days) versus a longer treatment (21days) in treating a first episode of probably idiopathic acute pericarditis. It is a non inferiority trial.

Exclusion criteria are: diseases known to cause pericarditis: (recent myocardial infarction, autoimmune disease, postpericardiotomy syndromes, connective tissue disease, tuberculosis, neoplastic disease).

Primary endpoint is: 30 days recovery defined as the normalization of all clinical and paraclinical initial abnormalities.

Secondary endpoint is: 6-month recurrence.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* first episode of acute pericarditis
* chest pain lasting less than 24 hours

Exclusion Criteria:

* contraindication to aspirin
* previous history of atypical chest pain
* previous history of connective tissue disease, tuberculosis, recent MI, auto immune disease, neoplastic disease, thoracic trauma, previous thoracic surgery, antiplatelet routine treatment, anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
recovery | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: jean-christophe cornily, md, Principal Investigator — FESC, Fellow of the french society of cardiology
Locations (12):
- France (12):
  - CHU de Brest, Brest
  - HIA Clermont Tonnerre, Brest
  - CHG Carhaix, Carhaix-Plouguer
  - CHG Douarnenez, Douarnenez
  - CH Lannion, Lannion
  - CHG Lorient, Lorient
  - Hôpital de la Timone, Marseille
  - CH Morlaix, Morlaix
  - Hôpital Claude Bernard APHP, Paris
  - Centre Hospitalier Intercommunal de Cornouaille, Quimper
  - CHG Saint-Brieuc, Saint-Brieuc
  - HIA Sainte-Anne, Toulon

REFERENCES:
- [Background] Maisch B, Seferovic PM, Ristic AD, Erbel R, Rienmuller R, Adler Y, Tomkowski WZ, Thiene G, Yacoub MH; Grupo de Trabajo para el Diagnostico y Tratamiento de las Enfermedades del Pericardio de la Sociedad Europea de Cardiologia. [Guidelines on the diagnosis and management of pericardial diseases. Executive summary]. Rev Esp Cardiol. 2004 Nov;57(11):1090-114. doi: 10.1016/s0300-8932(04)77245-0. No abstract available. Spanish. PMID 15544758
- [Background] Imazio M, Bobbio M, Cecchi E, Demarie D, Demichelis B, Pomari F, Moratti M, Gaschino G, Giammaria M, Ghisio A, Belli R, Trinchero R. Colchicine in addition to conventional therapy for acute pericarditis: results of the COlchicine for acute PEricarditis (COPE) trial. Circulation. 2005 Sep 27;112(13):2012-6. doi: 10.1161/CIRCULATIONAHA.105.542738. PMID 16186437